CLINICAL TRIAL: NCT04971668
Title: Effect of Aromatherapy Versus Gum Chewing on Preoperative Anxiety in Females Undergoing Gynecological Laparoscopy: A Randomized Controlled Trial
Brief Title: Aromatherapy Versus Gum Chewing on Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300635
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy; Chewing Gum; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy (Experimental): Designated blend aromatherapy (ginger & lavender) and patient will be asked to inhale deeply and simulate like chewing gum for 5 minutes.
  Interventions: Other: Aromatherapy
- Gum Chewing (Experimental): Patients will chew gum (sugar free) and inhale deeply with inert gauze for 5 minutes.
  Interventions: Other: Gum Chewing
- Placebo (Other): Patient will simulate like chewing gum and inhale deeply with inert gauze for 5 minutes.
  Interventions: Other: Controlled

INTERVENTIONS:
Other: Aromatherapy — Three drops of the designated blend aromatherapy (ginger & lavender) will be placed on a 2-inch by 2-inch impermeable, backed gauze pad and patient will be asked to inhale deeply and simulate like chewing gum for 5 minutes.
  Arms: Aromatherapy
Other: Gum Chewing — Patients will chew gum (sugar free) and inhale deeply with inert gauze for 5 minutes.
  Arms: Gum Chewing
Other: Controlled — Patients will inhale deeply with inert gauze and simulate like chewing gum for 5 minutes.
  Arms: Placebo

SUMMARY:
Investigators hypothesized that the use of blend aromatherapy and gum chewing before surgery would reduce preoperative anxiety as assessed by the Speilberger State-Trait Anxiety Inventory (STAI) questionnaire and provide non pharmacological methods to decrease postoperative sore throat, postoperative nausea & vomiting and postoperative pain.

DETAILED DESCRIPTION:
A written informed consent will be taken from the patients.patients will be assigned randomly to three groups (30 subjects each) either with preoperative aromatherapy (Group A) or gum chewing (Group G) or control group (Group C) to assess the preoperative anxiety and postoperative sore throat, nausea & vomiting and pain control between the three studied groups.

ELIGIBILITY:
Inclusion Criteria:

* Educated adult females
* American Society of Anesthesiologists (ASA) physical status I-II
* Listed for elective gynecological laparoscopy surgery under general anesthesia and endotracheal tube (ETT)

Exclusion Criteria:

* Impaired pharyngeal or esophageal function
* Phenylketonuria (contraindication to the sweetener aspartame in chewing gum)
* A fall upper or lower denture (not feasible to chew gum)
* A history of preoperative sore throat, upper respiratory tract illness
* Using steroid or analgesia within the last 48 hour
* Chronic smokers
* Receiving warfarin, heparin, full dose 325 mg aspirin, or clopidogrel
* A history or diagnosis of bleeding diatheses
* Any known allergies to ginger or lavender
* Having head or neck surgery
* History of difficult intubation
* Pregnant women

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety scale assessed by STAI questionnaire | Preoperative 15 minutes
  The STAI takes less than 5 minutes to complete and can be scored in less than 2 minutes. There are 20 questions (I feel calm, secure, tense, strained, at ease, upset, am presently worrying over possible misfortunes, satisfied, frightened, uncomfortable, self-confident, nervous, jittery, indecisive, relaxed, content, worried, confused, steady and pleasant) where people rate their anxiety from one (not at all) to four (very much so), and scores range from 20 to 80. For example, low anxiety is 20 to 37, moderate anxiety is 38 to 44, and high anxiety is 45 to 80. Assessment will be done at two times; first time (before study intervention)15 minutes preoperatively in the holding area as a baseline with recoding systolic blood pressure, diastolic blood pressure, heart rate and respiratory rate. Second time; (after study intervention) in the operating room before induction of anesthesia

SECONDARY OUTCOMES:
Postoperative sore throat (POST) score | Postoperative 24 hour
  On arrival in the post anesthesia care unit, the patient is immediately evaluated for the presence of postoperative sore throat (POST); time 0 hour using a standardized scale. The severity of POST is graded on a 4-point scale ranging from 0 to 3; 0 being no sore throat, 1 being mild discomfort (complains only with questioning), 2 being moderate sore throat (complains on their own), and 3 being severe sore throat (change in voice, hoarseness, and throat pain). Evaluations will be recorded at 0, 1, 2, 4, 6, 12 and 24 hours after surgery. Patients with score ≥2; will be given dexamethasone 4 mg and parecoxib 40 mg.
Postoperative nausea and vomiting (PONV) score | Postoperative 24 hour
  The post anesthesia care unit (PACU) nurses will assess and document postoperative nausea and vomiting (PONV) using a Verbal Descriptive Scale, which correlates to visual analog nausea scores, with an objective measure of severity: 0 = no PONV: patient reports no nausea and has had no emesis episodes; 1 = mild PONV: patient reports nausea but declines antiemetic treatment; 2 = moderate PONV: patient reports nausea and accepts antiemetic treatment; and 3 = severe PONV: nausea with any emesis episode (retching or vomiting). The score will be obtained at 0, 1, 2, 4, 6, 12 and 24 hours after PACU arrival. In the PACU, ondansetron 4 mg IV will be given for score ≥2.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Soliman, MD, Study Director — Omar makram
Locations (1):
- Assiut university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026